CLINICAL TRIAL: NCT06781060
Title: Effect of Faradic Nerve Stimulation on Post-Injection Sciatic Nerve Injury Pediatric Patients
Brief Title: Effect of Nerve Stimulation on Sciatic Nerve Injury Pediatric Patients
Acronym: PISNI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azeem Hospital, Multan (Other)
Responsible Party: Principal Investigator, Dr Chaman Lal, Physiotherapist, Azeem Hospital, Multan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AzeemH-01/MN/2024
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Leg Pain; Peripheral Nerve Discontinuities; Muscle Weakness; Sciatic Nerve Compression
Keywords: PISNI; FNS; ES; Peripheral Nerve Injury; Sciatic Nerve Traumatic Injury
MeSH Terms: conditions — Muscle Weakness; Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: The study outlined follows a randomized controlled trial (RCT) interventional model designed to assess the effectiveness of Faradic Nerve Stimulation (FNS) combined with standard physiotherapy in treating Post-Injection Sciatic Nerve Injury (PISNI) in pediatric patients. PISNI is a condition that typically occurs after an improper intramuscular (IM) injection, often leading to severe long-term consequences such as chronic pain, muscle weakness, and significant loss of mobility. While traditional treatment strategies, especially physiotherapy, are often used to manage PISNI, they may not always result in complete recovery. The primary aim of this study is to investigate whether the addition of FNS to standard physiotherapy could offer superior therapeutic benefits by improving nerve regeneration, alleviating pain, and enhancing functional mobility in children suffering from this injury.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faradic Nerve Stimulation Intervention Group A (Experimental): This is an intervention group in which Standard Physiotherapy + Electrical Nerve Stimulation will be provided to the participants.
  Interventions: Device: Faradic Nerve Stimulation Therapy+Standard Physiotherapy
- Control TENS Stimulation Group B (Active Comparator): This is control group in which Standard Physiotherapy + TENS Stimulation will be provided to the participants.
  Interventions: Device: Physiotherapy Standard Treatment with TENS machine therapy

INTERVENTIONS:
Device: Faradic Nerve Stimulation Therapy+Standard Physiotherapy — This is electrical nerve stimulation with faradic type current to the injured nerve for conservative treatment of post injection sciatic nerve injury.
  Arms: Faradic Nerve Stimulation Intervention Group A
Device: Physiotherapy Standard Treatment with TENS machine therapy — The control group in which Standard Physiotherapy + TENS therapy will be provided to the participants.
  Arms: Control TENS Stimulation Group B

SUMMARY:
Brief Summary The goal of this study is to learn if Faradic Nerve Stimulation (FNS) can help children recover from a condition called Post-Injection Sciatic Nerve Injury (PISNI). PISNI happens when the sciatic nerve, which controls muscles and sensation in the legs, gets injured from an injection that was given in the wrong place or in the wrong way. This injury can cause pain, muscle weakness, and problems moving the legs.

The main questions this study aims to answer are:

Can Faradic Nerve Stimulation help children with PISNI recover better than regular physiotherapy alone? Does FNS reduce pain and improve movement in children with this injury? What will happen in the study?

Children with PISNI will be treated in one of two groups:

Group A will receive Faradic Nerve Stimulation along with regular physiotherapy.

Group B will receive only regular physiotherapy and a similar treatment called Transcutaneous Electrical Nerve Stimulation (TENS).

Both treatments will be given by healthcare professionals in a safe and comfortable environment. Participants will be asked to attend therapy sessions for a few months and will be checked regularly to see how well they are recovering.

Why is this study important?

Post-Injection Sciatic Nerve Injury is common in children, especially in countries where healthcare providers may not be properly trained. This can lead to long-term problems, including pain and difficulty walking. Standard physiotherapy helps but doesn't always work well enough. By testing Faradic Nerve Stimulation, this study hopes to find a treatment that helps nerves heal faster and more completely, especially in children who need it most.

The findings from this study could lead to better treatments for nerve injuries in children, particularly in areas where healthcare resources are limited. If FNS works well, it could be a new way to help children recover and live pain-free lives.

DETAILED DESCRIPTION:
Background and Clinical Significance

Post-Injection Sciatic Nerve Injury (PISNI) is an important medical concern, particularly in children who are more vulnerable to this complication due to their developing anatomy and physiology. PISNI occurs when the sciatic nerve, which is responsible for motor and sensory functions in the lower limbs, is damaged during an intramuscular (IM) injection. This injury can result from improper needle placement, improper injection techniques, or repeated injections into the same site. PISNI leads to long-term disabilities including pain, muscle weakness, impaired mobility, and permanent nerve damage if not treated adequately. The prevalence of PISNI is notably higher in low-resource settings, where healthcare providers may lack proper training or access to necessary medical tools.

In Pakistan, studies have shown that the incidence of PISNI in pediatric populations ranges between 3.38% and 9%, primarily due to unsafe injection practices. Children in rural areas are especially at risk due to the limited availability of skilled healthcare providers, contributing to the increased occurrence of nerve injuries from IM injections. The repercussions of these injuries are not only physical but also emotional and social, as children face difficulties in performing everyday tasks and experience chronic pain, which can significantly reduce their quality of life.

Current treatment options for PISNI are limited, with most therapies focusing on pain relief and symptom management rather than promoting true nerve recovery or healing. Conventional physiotherapy has shown some benefit but is not always sufficient for complete recovery, especially in severe cases. Therefore, this study seeks to investigate the effectiveness of Faradic Nerve Stimulation (FNS) in treating PISNI and improving the recovery outcomes in pediatric patients.

The Proposed Solution: Faradic Nerve Stimulation (FNS) Faradic Nerve Stimulation (FNS) is an innovative therapeutic approach that uses low-frequency electrical pulses to stimulate muscles, improve nerve conduction, and promote nerve regeneration. The technique has been widely studied in the context of adult neuromuscular rehabilitation but remains underexplored in pediatric cases, particularly for PISNI. By stimulating the sciatic nerve and the surrounding muscles, FNS aims to enhance neuromuscular recovery, improve muscle strength, and reduce pain and inflammation.

FNS works by using a specific type of electrical current, typically of low frequency, to induce muscle contractions. These contractions help prevent muscle atrophy, enhance blood flow, and stimulate the regeneration of nerve fibers. Recent studies have suggested that FNS can promote neuroplasticity - the brain's ability to reorganize and form new neural connections - which may be critical in helping children recover from nerve injuries. Importantly, FNS provides a non-invasive, low-cost, and potentially scalable solution that can be applied even in low-resource settings, making it a promising adjunct therapy for PISNI.

The effectiveness of FNS compared to traditional physiotherapy has been the subject of some research, but few studies have focused on its use in pediatric populations with PISNI. This gap in the literature underscores the need for this study, which aims to compare the outcomes of FNS combined with standard physiotherapy versus standard physiotherapy alone.

Primary and Secondary Objectives The primary aim of this study is to evaluate the effectiveness of combining Faradic Nerve Stimulation with standard physiotherapy in the recovery of pediatric patients with Post-Injection Sciatic Nerve Injury (PISNI). The study will assess several key outcomes to determine if FNS offers additional benefits over conventional physiotherapy treatments.

Primary Objective

The primary objective is to evaluate and compare the electrophysiological recovery of sciatic nerve function in pediatric patients with PISNI treated with standard physiotherapy versus those treated with both standard physiotherapy and Faradic Nerve Stimulation. Specifically, the study aims to assess:

The impact of FNS on nerve conduction velocity and overall nerve regeneration in children with PISNI.

The potential improvement in muscle strength and motor function. Secondary Objectives

In addition to the primary objective, the study also seeks to evaluate the broader effects of combining FNS with physiotherapy, including:

Pain Reduction: Assessing whether FNS reduces pain intensity compared to physiotherapy alone.

Functional Mobility: Evaluating improvements in the ability of children to move and perform daily activities as measured by functional mobility scales.

Quality of Life (QOL): Measuring the impact on the family's well-being and the child's quality of life using validated questionnaires.

Study Design and Methodology

This study is designed as a Randomized Controlled Trial (RCT), which is widely considered the gold standard for evaluating the effectiveness of medical interventions. A total of 80 pediatric patients, aged between 3 and 19 years, who have been diagnosed with PISNI, will be recruited for this study. The participants will be randomly allocated into two groups:

Group A (Intervention Group): This group will receive Faradic Nerve Stimulation combined with standard physiotherapy.

Group B (Control Group): This group will receive standard physiotherapy along with Transcutaneous Electrical Nerve Stimulation (TENS), another common electrical stimulation therapy.

Group A will receive Faradic Nerve Stimulation along with standard physiotherapy. FNS will be applied using low-frequency electrical pulses, targeting the sciatic nerve and the affected muscles.

Group B will receive TENS along with standard physiotherapy. TENS uses electrical impulses to help manage pain by blocking pain signals and stimulating the release of endorphins.

Follow-Up Phase: After the treatment phase, both groups will be monitored for an additional 4 weeks to track any ongoing recovery or improvements. During this period, participants will undergo follow-up assessments to measure the sustainability of improvements in pain reduction, motor function, and quality of life.

Statistical Analysis The collected data will be analyzed using advanced statistical methods. ANOVA (Analysis of Variance) will be used for between-group comparisons, while paired t-tests will be employed to evaluate within-group changes over time. The study will also calculate effect sizes (Cohen's d > 0.8) to determine the clinical significance of the results.

Detailed Study Design: Participant Selection and Randomization Participant Recruitment and Screening The recruitment process will focus on identifying children aged 3 to 19 years who are diagnosed with Post-Injection Sciatic Nerve Injury (PISNI) caused by improper intramuscular (IM) injections. Pediatric participants will be recruited from tertiary care centers that manage PISNI cases. To ensure the robustness and validity of the findings, the study will employ a simple randomization method to allocate participants to either the intervention group (Group A) or the control group (Group B).

Before enrollment, each participant's eligibility will be verified through a thorough screening process. This will include confirming the diagnosis of PISNI, ensuring no other underlying health conditions that could influence treatment outcomes, and obtaining written consent from a parent or guardian for the child's participation. Given the potential for unqualified providers to administer injections, special attention will be given to the documentation and verification of the injury's origin to rule out non-iatrogenic causes of nerve injury.

Intervention Procedures Group A (Intervention Group): Faradic Nerve Stimulation (FNS) + Standard Physiotherapy The intervention group will receive a combination of Faradic Nerve Stimulation (FNS) and standard physiotherapy. FNS involves the application of low-frequency electrical impulses to stimulate neuromuscular recovery. The electrical pulses are delivered to the affected muscles and sciatic nerve through surface electrodes. The therapy aims to induce rhythmic muscle contractions that assist in preventing atrophy, improving muscle tone, and facilitating nerve regeneration.

FNS will be applied at specific frequencies (50-100 Hz) and pulse durations (0.1-1 milliseconds) to ensure effective stimulation without causing discomfort to the patient. Treatment sessions will be scheduled three times a week, lasting 20-30 minutes per session. Along with FNS, children will also receive standard physiotherapy interventions, including strength exercises, functional mobility training, and manual therapy, to improve muscle coordination and promote recovery.

Group B (Control Group): Standard Physiotherapy + Transcutaneous Electrical Nerve Stimulation (TENS)

The control group will receive standard physiotherapy treatment along with Transcutaneous Electrical Nerve Stimulation (TENS). TENS uses electrical impulses delivered through surface electrodes placed on the skin to reduce pain and discomfort. The mechanism of TENS involves stimulating sensory nerves and blocking pain signals from reaching the brain, helping to manage pain while allowing the body to heal.

TENS will be applied using frequencies between 2 Hz and 100 Hz, with pulse durations ranging from 50 to 250 microseconds. While TENS is effective for pain management, it does not promote nerve regeneration or motor recovery to the extent that FNS does. Therefore, the control group will also receive standard physiotherapy, which includes strengthening exercises and functional mobility training, similar to the intervention group.

Treatment Schedule:

Both groups will undergo therapy for 8 weeks and till16 weeks. Sessions will take place three times a week. Follow-up assessments will be conducted for 4 weeks after the treatment phase to monitor ongoing recovery.

Outcome Measures and Data Collection Primary Outcome: Electrophysiological Recovery

The primary outcome of this study is the electrophysiological recovery of the sciatic nerve. This will be assessed by measuring the nerve conduction velocity (NCV), which reflects the speed of electrical signals traveling through the nerve. Faster nerve conduction indicates improved nerve function and regeneration.

Secondary Outcomes:

Pain Management: Pain will be assessed using the Wong-Baker FACE Scale and the FLACC Pediatric Pain Scale, which measure pain intensity through facial expressions, body movements, and verbal cues in children.

Functional Mobility: The study will use the Pediatric Evaluation of Disability Inventory (PEDI), which assesses functional abilities in children, including self-care, mobility, and social function.

Quality of Life: The Pediatric Quality of Life Family Impact Module (PQL-FIM) will be used to evaluate the impact of PISNI on the child's quality of life and the well-being of their family.

Follow-Up Phase: Monitoring Recovery After the completion of the treatment phase, participants will enter the Follow-Up Phase, which lasts for 4 weeks. During this phase, children will be re-assessed to evaluate the sustainability of their recovery and improvements in functional mobility, pain levels, and overall quality of life. The follow-up phase will also help identify any delayed effects of treatment, which are common in nerve injuries.

The follow-up visits will be spaced at regular intervals to track recovery progress and ensure any complications are promptly addressed. All assessments will be conducted using the same standardized tools to allow for accurate comparisons to baseline measurements.

Statistical Analysis

Data Processing and Statistical Methods:

Data analysis will be performed using SPSS (Statistical Package for the Social Sciences) software. Descriptive statistics will be used to summarize the demographics of the participants, including age, gender, and baseline measurements of pain, mobility, and quality of life. The main data analysis methods will include:

Analysis of Variance (ANOVA): This will be used to compare the outcomes between the two groups at the end of the treatment phase. ANOVA will allow the researchers to assess whether the combination of FNS and physiotherapy significantly improves recovery outcomes compared to standard physiotherapy alone.

Paired t-tests: This will be used to compare within-group differences before and after the treatment period, which will help measure improvements over time for each group.

Effect Size Calculation: The study will calculate Cohen's d to determine the clinical significance of the results. An effect size of Cohen's d > 0.8 will be considered significant, indicating a large treatment effect.

Handling Missing Data:

In cases of missing data, the study will use imputation methods to estimate the missing values based on available data, ensuring the accuracy and validity of the findings. Exploratory Data Analysis (EDA) will be performed to identify any outliers or anomalies in the data, which will be addressed before conducting formal statistical analyses.

Ethical Considerations This study will be conducted in accordance with the Declaration of Helsinki on ethical principles for medical research. Prior to enrollment, written informed consent will be obtained from the parents or guardians of all participants. Additionally, assent will be sought from children, when applicable, depending on their age and ability to understand the nature of the study.

The research will adhere to strict confidentiality guidelines, ensuring that all personal health information is securely stored and only accessible to authorized research personnel. The study will also be conducted in compliance with local regulations and institutional review board (IRB) guidelines. Regular ethical reviews will be carried out to ensure the safety and well-being of participants throughout the study.

Study Limitations

While the study is designed to rigorously evaluate the effects of Faradic Nerve Stimulation in the treatment of PISNI, there are several limitations that need to be considered:

Generalizability: The study is limited to children with PISNI and may not be applicable to adults or other types of peripheral nerve injuries.

Selection Bias: As with any RCT, there is a risk of selection bias, particularly due to the inclusion and exclusion criteria. The results may not apply to children with severe cases of PISNI or those who have other neurological conditions.

Treatment Protocol Variability: While every effort will be made to standardize the treatment protocol, there could be variability in how the interventions are administered, depending on the healthcare provider or the participant's response to treatment.

Long-Term Effects: The study will follow participants for a relatively short period (16 weeks). Long-term effects of FNS on pediatric nerve injuries will need to be assessed in future studies with longer follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with Post-Injection Sciatic Nerve Injury (PISNI) caused by improper intramuscular (IM) injections.
* Children aged 3 to 19 years.
* Parental consent for participation in the study.
* Assent from the child (when applicable), depending on the age and understanding of the participant.

Exclusion Criteria:

* Children requiring surgical intervention for severe neurotmesis.
* Patients with neurological or musculoskeletal conditions that may affect the outcomes (e.g., muscular dystrophy, multiple sclerosis).
* Children who are unable to participate in physical therapy due to other medical conditions or severe limitations.
* Children with severe systemic or other comorbid conditions that could interfere with study participation or outcome measures.

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Nerve Conduction Study (NCS) | The primary outcome will be assessed at baseline (pre-treatment) and at the end of the 8-week and final at 16 weeks treatment phase, to monitor ongoing recovery.
  The primary outcome measure evaluates the electrophysiological recovery of the sciatic nerve in pediatric participants with Post-Injection Sciatic Nerve Injury (PISNI). This is assessed through nerve conduction velocity (NCV), latency & amplitude, which measures the speed of electrical signals traveling through the sciatic nerve. An improvement in NCV indicates successful nerve regeneration and recovery of nerve function. The outcome will compare participants receiving Faradic Nerve Stimulation (FNS) combined with standard physiotherapy to those receiving Transcutaneous Electrical Nerve Stimulation (TENS) with standard physiotherapy.

SECONDARY OUTCOMES:
FLACC Pediatric Pain Scale | At Baseline, 8 weeks and 16 weeks
  Rates pain based on observable behaviors like facial expressions, leg movement, and crying. It provides ranked scores but without equal intervals.
Wong-Baker FACES Pain Scale | At Baseline, 8 weeks and 16 weeks
  Subjects rate their pain using facial expressions representing varying levels of discomfort, arranged in a ranked order.
Pediatric Quality of Life Family Impact Module (PQL-FIM) | The primary outcome will be assessed at baseline (pre-treatment) and at the end of the 8-week and final at 16 weeks treatment phase, to monitor ongoing recovery.
  The primary outcome measure assesses the improvement in quality of life of pediatric participants with Post-Injection Sciatic Nerve Injury (PISNI). This will be measured using the Pediatric Quality of Life Family Impact Module (PQL-FIM), which evaluates the impact of the child's health condition on the child's quality of life as well as the well-being of their family. Improvements in scores indicate a positive change in the child's daily functioning and family well-being.
  The PQL-FIM tool will be used to assess the quality of life in both groups (those receiving Faradic Nerve Stimulation (FNS) with physiotherapy and those receiving Transcutaneous Electrical Nerve Stimulation (TENS) with physiotherapy).
Pediatric Evaluation of Disability Inventory (PEDI) | The primary outcome will be assessed at baseline (pre-treatment) and at the end of the 8-week and final at 16 weeks treatment phase, to monitor ongoing recovery.
  The primary outcome measure evaluates the improvement in functional mobility in pediatric participants with Post-Injection Sciatic Nerve Injury (PISNI). This will be measured using the Pediatric Evaluation of Disability Inventory (PEDI), which assesses a child's ability to perform self-care, mobility, and social function. An improvement in functional mobility scores will indicate better recovery of physical abilities and independence. The measure will compare the outcomes between participants receiving Faradic Nerve Stimulation (FNS) combined with standard physiotherapy and those receiving Transcutaneous Electrical Nerve Stimulation (TENS) with physiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr Muhammad Zia Ul Haq Professor-Supervisor, PhD, Study Director — Lincoln University College (LUC), Malaysia
Locations (1):
- Azeem Hospital Mutan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study team plans to share individual participant data (IPD) with other researchers upon request. This will include de-identified data related to the primary and secondary outcome measures, including nerve conduction velocity, pain intensity scores, functional mobility assessments, and quality of life evaluations. The data will be made available in accordance with ethical guidelines, ensuring participant confidentiality and privacy. Data sharing will be facilitated through a secure platform, and only authorized researchers will be granted access to the dataset for further analysis. Requests for access to the data will be reviewed by the study's ethics committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after completion of the study and final statistical analysis. It will be available for researchers for 3 years after the completion of the study.
Access Criteria: The approved researchers, including academic institutions, healthcare professionals, and research organizations, who have a legitimate research interest and have received ethical approval to access the data, will be able to access the IPD and supporting information.
  Researchers will be able to access de-identified individual participant data (IPD), including nerve conduction velocity (NCV), pain intensity scores, functional mobility assessments, and quality of life data.
  Access to the data and supporting information will be provided through a secure online platform. Researchers will need to submit a formal request outlining the purpose of the data use. The request will be reviewed and approved by the study's ethics committee to ensure compliance with privacy regulations and ethical guidelines. Once approved, access will be granted to the appropriate data, and researchers will be required to adhere to confidentiality agreements and data protection standards.